CLINICAL TRIAL: NCT05464771
Title: The Impact of Patient Safety Incidents on Patients' Quality of Life
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 123
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Hip Fractures; Knee Fracture
MeSH Terms: conditions — Hip Fractures; Knee Fractures | interventions — Surgical Procedures, Operative; Papaverine; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients experiencing adverse event while in hospital: Patients that have experienced a patient safety incident according to the Patient Safety Indicators (PSIs) developed by the U.S. Agency for Healthcare Research and Quality (AHRQ)
  Interventions: Procedure: Surgery for hip and knee replacement

INTERVENTIONS:
Procedure: Surgery for hip and knee replacement — Elective inpatient surgery for hip and knee replacement

SUMMARY:
This study estimates the impact of patient safety events on QoL in elective surgery patients using a secondary data set

DETAILED DESCRIPTION:
Background: The burden of patient safety incidents (PSIs) is often characterised by their impact on mortality, morbidity and treatment costs. Few studies have attempted to estimate the impact of PSIs on patients' health-related quality of life (HRQoL) and the studies that have made such estimates primarily focus on a narrow set of incidents. The aim of this paper is to estimate the impact of PSIs on HRQoL of patients undergoing elective surgery in England.

Materials and Methods: A unique linked longitudinal data set consisting of Patient Reported Outcome Measures (PROMS) for patients with hip and knee replacements linked to Hospital Episode Statistics (HES) collected between 2013/14 and 2016/17 is examined. Patients with any of nine US Agency for Healthcare Research and Quality (AHRQ) PSI indicators are identified. HRQoL is measured using the general EuroQol five dimensions questionnaire (EQ-5D) before and after surgery. Exploiting the longitudinal structure of the data, exact matching combined with difference in differences to estimate the impact of experiencing a PSI on HRQoL and its individual dimensions, comparing HRQoL improvements after surgery in similar patients with and without a PSI.

ELIGIBILITY:
Inclusion Criteria:

* no

Exclusion Criteria:

* Patients for which health related quality of life is not observed both before and after surgery.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The data available for our study was collected between 2013 and 2017. The patient safety incidents studied are relatively rare, and in order to yield enough observations to reliably estimate the impact of different incidents, the sample is limited to patients undergoing hip or knee replacements because these have more observations than do varicose veins and groin hernia. There are 267,477 and 288,967 observations for patients undergoing hip replacement and knee replacement respectively. Furthermore, the sample is limited to patients with observations of health status both before and after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 395346 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
EuroQual - 5 Dimensions (EQ5D) | 2013-17
  quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Acute Trusts in England, Multiple Locations, United Kingdom

REFERENCES:
- [Derived] Xiao M, Kristensen SR, Marti J, Mossialos E. The impact of patient safety incidents during hip and knee replacements on patients' health related quality of life: a before and after study using longitudinal data linked to patient-reported outcome measures. Int J Surg. 2023 May 1;109(5):1085-1093. doi: 10.1097/JS9.0000000000000275. PMID 37026831